CLINICAL TRIAL: NCT01425632
Title: A Confirmatory Study of TAU-284 in Pediatric Patients With Perennial Allergic Rhinitis (A Randomized, Double-blind, Placebo-controlled Study)
Brief Title: A Confirmatory Study of TAU-284 in Pediatric Patients With Perennial Allergic Rhinitis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Tanabe Pharma Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: TAU-284-17
Record Dates: First submitted 2011-08-28; First posted 2011-08-30 (Estimated); Results first posted 2015-12-14 (Estimated); Last update posted 2026-01-07 (Actual); Status verified 2025-12

CONDITIONS: Perennial Allergic Rhinitis
Keywords: TAU-284; Bepotastine besilate; Histamine H1 receptor antagonists
MeSH Terms: conditions — Rhinitis, Allergic, Perennial | interventions — bepotastine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- TAU-284 Low (Experimental)
  Interventions: Drug: TAU-284
- TAU-284 High (Experimental)
  Interventions: Drug: TAU-284
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: TAU-284 — TAU-284 Low
  Arms: TAU-284 Low
Drug: TAU-284 — TAU-284 High
  Arms: TAU-284 High
Drug: Placebo — Placebo
  Arms: Placebo

SUMMARY:
The objectives of this study are: to confirm the superiority of TAU-284 over placebo after two weeks of administration to pediatric patients with perennial allergic rhinitis, and to investigate the dose response, safety, and plasma concentrations of TAU-284.

DETAILED DESCRIPTION:
This is a randomized, double-blind, placebo-controlled, 3-arm parallel-group comparative study to confirm the superiority of TAU-284 over placebo after two weeks of administration of TAU-284 (10 mg/day or 20 mg/day) or placebo to pediatric patients with perennial allergic rhinitis, with "the change from baseline in total nasal symptom score (total score for the three major nasal symptoms [sneezing, rhinorrhea, and nasal congestion])" as the primary endpoint; and to investigate the dose response, safety, and plasma concentrations of TAU-284.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged between 7 and 15 years
* Patients with a weight of at least 20 kg
* Patients who have received a diagnosis of perennial allergic rhinitis according to the diagnostic criteria
* Patients with a mean rhinorrhea score of at least 2 and a mean total score for the three major nasal symptoms [sneezing, rhinorrhea, and nasal congestion] of at least 4 on the basis of symptoms recorded in the nasal allergy diary during the observation period

Exclusion Criteria:

* Patients with vasomotor rhinitis or eosinophilic rhinitis
* Patients who have concurrent nasal disease that may affect the efficacy of TAU-284
* Patients with a history of any of the nasal surgical procedures
* Patients who have a positive result for pollen antigens which are dispersed during the study period
* Patients who have a positive result for dog dander or cat dander antigen
* Patients with current or previous history of drug allergy
* Patients who concurrently have renal function abnormalities that may cause safety problems

Ages: 7 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 490 (Actual)
Dates: Start 2011-08; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kimihiro Okubo, M.D. Ph.D., Study Director — Department of Otorhinolaryngology, Nippon Medical School
Locations (5):
- Japan (5):
  - Reserch site, Chūbu
  - Reserch site, Hokuriku
  - Reserch site, Kanto
  - Reserch site, Kinki
  - Reserch site, Kyusyu

RESULTS

PARTICIPANT FLOW:
Groups:
- TAU-284 Low: TAU-284 5mg twice daily for 2 weeks
- TAU-284 High: TAU-284 10mg twice daily for 2 weeks
- Placebo: TAU-284 placebo twice daily for 2 weeks
Period: Overall Study
Arm/Group | TAU-284 Low | TAU-284 High | Placebo
Started | 161 | 166 | 163
Completed | 160 | 165 | 159
Not Completed | 1 | 1 | 4
Not completed — Adverse Event | 0 | 1 | 1
Not completed — Physician Decision | 1 | 0 | 0
Not completed — Protocol Violation | 0 | 0 | 2
Not completed — Withdrawal by Subject | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | TAU-284 Low | TAU-284 High | Placebo | Total
Number analyzed (Participants) | 161 | 166 | 163 | 490
Age, Continuous [Mean (Standard Deviation); unit: years] | 11.2 (2.5) | 11.4 (2.3) | 11.2 (2.5) | 11.2 (2.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 62 | 64 | 72 | 198
  Male | 99 | 102 | 91 | 292

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Total Score for the Three Major Nasal Symptoms [Sneezing, Rhinorrhea, and Nasal Congestion] (at Final Evaluation)
Description: Total score for the three major nasal symptoms (sneezing, rhinorrhea, and nasal congestion) were rated on 4-point scale ranging from 0 (no symptoms) to 3 (severe) .
Time Frame: Baseline and Week 2
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | TAU-284 Low | TAU-284 High | Placebo
Number analyzed (Participants) | 161 | 166 | 163
units on a scale | -0.84 (0.12) | -0.92 (0.12) | -0.70 (0.12)

2. Secondary Outcome: Change From Baseline in Total Score for the Three Major Nasal Symptoms [Sneezing, Rhinorrhea, and Nasal Congestion]
Time Frame: Week 2
Reporting Status: Not Posted

3. Secondary Outcome: Change From Baseline in Individual Nasal Symptom Scores (Sneezing, Rhinorrhea, Nasal Congestion, and Impairment in Daily Activities)
Time Frame: Week 2
Reporting Status: Not Posted

4. Secondary Outcome: Change From Baseline in Individual Scores for Local Nasal Findings (Rhinoscopic Findings)
Time Frame: Week 2
Reporting Status: Not Posted

5. Secondary Outcome: Change From Baseline in Severity Score
Time Frame: Week 2
Reporting Status: Not Posted

6. Secondary Outcome: Adverse Events and Adverse Drug Reactions
Time Frame: Week 2
Reporting Status: Not Posted

7. Secondary Outcome: Plasma Concentrations of Unchanged TAU-284 (Bepotastine Besilate) (at a Total of 3 Time Points, i.e., Before and 2 (±1) Hours After Study-drug Administration at Week 1 and Before Study-drug Administration at Week 2)
Time Frame: Week 2
Reporting Status: Not Posted

ADVERSE EVENTS:
Arm/Group | TAU-284 Low | TAU-284 High | Placebo
Serious Adverse Events (participants affected / at risk) | 0/161 | 0/166 | 0/163
Other Adverse Events (participants affected / at risk) | 17/161 | 8/166 | 15/163
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | TAU-284 Low (N=161) | TAU-284 High (N=166) | Placebo (N=163)
Nasopharyngitis (Infections and infestations) | 8 | 3 | 11
Pharyngitis (Infections and infestations) | 5 | 2 | 4
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 5 | 4 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other